CLINICAL TRIAL: NCT04013646
Title: Safety and Efficacy of Combined Administration of Erythropoietin in Umbilical Cord Blood Therapy for Stroke Patients
Brief Title: Combination Therapy of Umbilical Cord Blood and Erythropoietin for Stroke Paients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bundang CHA Hospital (Other)
Collaborators: Korea Evaluation Institute of Industrial Technology (Other)
Responsible Party: Principal Investigator, MinYoung Kim, MD, PhD, Head of Rehabilitation Medicine Department, Professor, Principal Investigator, Bundang CHA Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018-12-030
Record Dates: First submitted 2019-07-08; First posted 2019-07-10 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Stroke; Umbilical Cord Blood; Erythropoietin; Safety; Treatment Outcome
MeSH Terms: conditions — Stroke | interventions — Erythropoietin; Rehabilitation

STUDY DESIGN:
Intervention Model Description: Group 1: UCB infusion and EPO injection group Group 2: UCB infusion and placebo EPO injection group Group 3: Placebo UCB infusion and placebo EPO injection group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- UCB infusion and EPO injection group (Experimental): Take immunosuppressant agents for 1 week. Umbilical cord blood is administered in the treatment room. Afterward, the venous erythropoietin agent injects into the peripheral vein 5 times a total of 5 times a week.
  Interventions: Drug: Placebo umbilical cord blood infusion; Drug: Placebo erythropoietin injection; Procedure: Active rehabilitation
- UCB infusion and placebo EPO injection group (Experimental): Take immunosuppressant agents for 1 week. Umbilical cord blood is administered in the treatment room. Afterward, the venous erythropoietin placebo injects into the peripheral vein 5 times a total of 5 times a week.
  Interventions: Drug: Umbilical cord blood infusion; Drug: Placebo erythropoietin injection; Procedure: Active rehabilitation
- Placebo UCB infusion and placebo EPO injection group (Placebo Comparator): Take immunosuppressant placebo for 1 week with the same schedule as the experimental group. As in the experimental group, placebo umbilical cord blood is administered in the treatment room and stay in the treatment room for the same time. Afterward, the venous erythropoietin placebo injects into the peripheral vein 5 times a total of 5 times a week. Other inspection schedules proceed with other groups.
  Interventions: Drug: Umbilical cord blood infusion; Drug: Erythropoietin injection; Procedure: Active rehabilitation

INTERVENTIONS:
Drug: Umbilical cord blood infusion — The umbilical cord blood is donated umbilical cord blood which is stored in the cord blood bank donated by Cha Hospital. The total number of nuclear cells should be at least 2 x 10 7 / kg, and at least three out of six of the six human leukocyte antigens (HLA-A, B, DR) should be selected. The cord blood that matches ABO and Rh blood type is preferentially used. Umbilical cord blood infusion is administered intravenously and is performed at the stem cell clinical trial center. The procedure is performed by the doctor who is enrolled in this study. Monitor pulse and oxygen saturation during the procedure.
  Other Names: UCB
  Arms: Placebo UCB infusion and placebo EPO injection group; UCB infusion and placebo EPO injection group
Drug: Erythropoietin injection — Recombinant human erythropoietin is used and is administered intravenously at a maximum of 5 times at a rate of 500 IU / kg 2 times/week after cord blood peripheral blood infusion, calculated as the dose per body weight. Or subcutaneous administration if intravenous administration is not possible. Store in a sealed container at 2-8 °C in the refrigerator before dosing. Erythropoietin injection is performed at the stem cell clinical trial center. The procedure is performed by the doctor who is enrolled in this study. Monitor pulse and oxygen saturation during the procedure.
  Other Names: EPO
  Arms: Placebo UCB infusion and placebo EPO injection group
Drug: Placebo umbilical cord blood infusion — Placebo umbilical cord blood infusion is administered intravenously and is performed at the stem cell clinical trial center. The procedure is performed by the doctor who is enrolled in this study. Monitor pulse and oxygen saturation during the procedure.
  Other Names: pUCB
  Arms: UCB infusion and EPO injection group
Drug: Placebo erythropoietin injection — Placebo erythropoietin injection is performed at the stem cell clinical trial center. The procedure is performed by the doctor who is enrolled in this study. Monitor pulse and oxygen saturation during the procedure.
  Other Names: pEPO
  Arms: UCB infusion and EPO injection group; UCB infusion and placebo EPO injection group
Procedure: Active rehabilitation — Physical therapy and occupational therapy are performed daily.
  Other Names: Rehabilitation

SUMMARY:
This clinical trial is a clinical trial for the evaluation of the safety and efficacy of umbilical cord blood (UCB) therapy, UCB and erythropoietin (EPO) combination therapy in adult stroke patients.

DETAILED DESCRIPTION:
UCB is a high-quality source of mesenchymal stem cells, and studies are being actively developed for stroke patients. UCB therapy has a neuroprotective effect through anti-inflammatory effect and anti-apoptosis.

However, UCB alone has not been able to provide sufficient improvement and is being studied for combination therapies with growth factors that can exert its effects. Among the various growth factors, EPO is a powerful factor that can act as a neurotrophic factor in neurons, astrocytes, oligodendrocytes, microglia, endothelial cells, and neural stem/precursor cells.

In our previous study of subacute stroke animal models, investigators confirmed that the combined administration of UCB and EPO improved the behavioral assessment (mNSS, Cylinder test) compared to UCB only administration.

The aim of this study is to investigate the difference in therapeutic effects between UCB alone therapy and UCB and EPO combination therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients over 20 years old
2. Patients with a stroke lasting from 30 days to less than 9 months
3. After hearing and fully understanding the details of this clinical trial, the person or legal representative has agreed to voluntary participation and has agreed in writing to comply with the notice

Exclusion Criteria:

Patients with one or more of the following can not participate in the study.

1. Patients with uncontrolled hypertension
2. A person who has impaired ability of consent, who is not accompanied by a guardian
3. Women who are pregnant, lactating, have a pregnancy plan during the trial, or those who do not use an available contraceptive method (women of childbearing age must be negative in the pregnancy test on baseline visit (0 weeks) .)
4. Those who satisfy the following conditions

   * A person whose ALT / AST is measured at 120 IU / L or more
   * Serum creatinine greater than 1.8 mg / dL
   * Total bilirubin> 1.8 mg / dL
   * Total WBC count less than 3000 / mm3
   * Those with a Hb of 16 g / dL or more
   * Platelet count less than 150,000 / uL or more than 675,000 / uL
5. Clinically significant infections during the screening period (pneumonia, pyelonephritis, sepsis, etc.)
6. Persons with severe medical conditions such as cardiovascular, digestive, respiratory, and endocrine conditions.
7. Any kind of confirmed congenital or acquired immune deficiency syndrome
8. Those who have been diagnosed with malignant carcinoma (excluding complete remission for more than 10 years)
9. If participants have side effects on your medication [Regarding erythropoietin agent]

   * Patients with hypersensitivity to erythropoietin
   * Patients sensitive to mammalian cell-derived drugs or human albumin
   * epileptic patients
   * Patients with a history of seizures
   * Patients on a thrombolytic drug (meaning thrombolytic agent such as Tissue Plasminogen Activator, allowing anti-platelet agents such as aspirin and plavix) [Related to tacrolimus] Patients with hypersensitivity to tacrolimus or macrolide compounds
   * Patients receiving cyclosporine or bosentan
   * Patients receiving potassium-preserving diuretics
10. Other If the investigator determines that participation in this trial is not appropriate

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-05-02 (Actual); Primary Completion 2020-11-02 (Estimated); Study Completion 2021-11-02 (Estimated)

PRIMARY OUTCOMES:
Change of Functional Independence Measure | baseline - 3 months - 6 months
  The difference in the FIM (Functional Independence Measure)score between the three groups at baseline, 90 days, and 180 days was confirmed by comparing differences in scores (total score[18~126], motor score[13~90], and cognition score[5~35]. The total score is the sum of the motor score and the cognition score. The higher scores represent a better outcome )

SECONDARY OUTCOMES:
Change of Medical research council | baseline - 3 months - 6 months
  The difference in the MRC (Medical research council) scale between the three groups at baseline, 90 days, and 180 days was confirmed by comparing differences. [0, 1, 2, 2, 2+, 3-, 3, 3+, 4, 5] (The higher values represent a better outcome.)
Change of National Institutes of Health Stroke Scale | baseline - 3 months - 6 months
  The difference in the NIHSS (National Institutes of Health Stroke Scale) between the three groups at baseline, 90 days, and 180 days was confirmed by comparing differences.[0~42] (The lower values represent a better outcome.)
Change of Manual Function Test | baseline - 3 months - 6 months
  The difference in the MFT (Manual Function Test) between the three groups at baseline, 90 days, and 180 days was confirmed by comparing differences.[0~32 for each arm] (The higher values represent a better outcome.)
Change of Fugl-Meyer Assessment | baseline - 3 months - 6 months
  The difference in the FMA (Fugl-Meyer Assessment) between the three groups at baseline, 90 days, and 180 days was confirmed by comparing differences.[0~66 for each arm] (The higher values represent a better outcome.)
Change of Berg Balance Scale | baseline - 3 months - 6 months
  The difference in the BBS (Berg Balance Scale) between the three groups at baseline, 90 days, and 180 days was confirmed by comparing differences.[0~56] (The higher values represent a better outcome.)
Change of Trunk Imbalance Scale | baseline - 3 months - 6 months
  The difference in the TIS (Trunk Imbalance Scale) between the three groups at baseline, 90 days, and 180 days was confirmed by comparing differences.[0~23] (The higher values represent a better outcome.)
Change of Korean Mini Mental State Exam | baseline - 3 months - 6 months
  The difference in the K-MMSE (Korean Mini Mental State Exam) between the three groups at baseline, 90 days, and 180 days was confirmed by comparing differences. [0~30] (The higher values represent a better outcome.)
Change of Korean Wechsler adult intelligence scale-IV | baseline - 3 months - 6 months
  The difference in the K-WAIS-IV (Korean Wechsler adult intelligence scale-IV) between the three groups at baseline, 90 days, and 180 days was confirmed by comparing differences.[The total score is a standard score with a mean of 100 and a standard deviation of approximately 15.] (The higher values represent a better outcome.)
Change of Korean version of the Western Aphasia Battery | baseline - 3 months - 6 months
  The difference in the K-WAB (Korean version of the Western Aphasia Battery) between the three groups at baseline, 90 days, and 180 days was confirmed by comparing differences.[0~100] (The higher values represent a better outcome.)
Change of Brain imaging | baseline - 6 months
  The difference in the Brain imaging (Basic brain MRI, functional brain MRI, diffusion tensor imaging brain MRI) between the three groups at baseline, and 180 days was confirmed by comparing differences.
Change of Biomarkers | baseline - 1 day - 15 days - 1 month - 3 months - 6 months
  The difference in the Biomarkers (TGFβ, IL-10, IL-8, PTX3, PCNT,...) between the three groups at baseline, 1 day, 15 days, 30 days, 90 days and 180 days was confirmed by comparing differences.

CONTACTS AND LOCATIONS:
Overall Officials: MinYoung Kim, MD,PhD, Study Director — CHA Bundang Medical Center
Locations (1):
- Bundang CHA Medical Center, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim JM, Shin S, Lee D, Choi JI, Kwon HG, Hwang SSS, Cho SM, Kim YH, Lee J, Moon HI, Suh MR, Kim M. Safety and efficacy of allogeneic umbilical cord blood cells and erythropoietin combination therapy in patients with subacute stroke. Stem Cell Res Ther. 2025 Dec 27;17(1):56. doi: 10.1186/s13287-025-04856-8. PMID 41456040